CLINICAL TRIAL: NCT03387839
Title: Antero-Posterior Knee Stability With Medial-Pivot, Cruciate-Substituting, and Posterior-Stabilized Total Knee Arthroplasty: A Retrospective Study
Brief Title: Antero-Posterior Knee Stability
Status: Completed | Type: Observational
Sponsor: David F. Scott, MD (Other)
Responsible Party: Sponsor-Investigator, David F. Scott, MD, Principal Investigator, Spokane Joint Replacement Center
Organization: Spokane Joint Replacement Center (Other)
Other Study IDs: SJRC-AP-Stability
Record Dates: First submitted 2017-12-11; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis; Total Knee Arthroplasty; Stability; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (3):
- Medial-Pivot Knee Prosthesis
  Interventions: Other: Stress X-Ray
- Posterior-Stabilized Knee Prosthesis
  Interventions: Other: Stress X-Ray
- Cruciate-Stubstituting Knee Prosthesis
  Interventions: Other: Stress X-Ray

INTERVENTIONS:
Other: Stress X-Ray — Antero-posterior stability of the knee measured with stress x-rays using the TELOS Stress device in 45° and 90° flexion

SUMMARY:
A retrospective one-time evaluation of total knee patients one year or more postoperative, to compare antero-posterior (AP) stability with the TELOS Stress device/stress x-rays and clinical outcomes. Multiple implant brand/models will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign the informed consent.
* Patients able to comply with study requirements including stress x-rays and self-evaluations.
* Male and non-pregnant females ages 21 - 80 years of age at the time of surgery.
* Patients who have undergone a primary total knee replacement, are one year or greater postoperative, and are not having any evidence of failure of their implants.
* Patients with a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
* Patients with intact collateral ligaments.
* Range of motion within five degrees of full extension and a minimum of 120 degrees of flexion.

Exclusion Criteria:

* Patients with inflammatory arthritis.
* Patients that are morbidly obese, body mass index (BMI) > 40.
* Patients that have had a high tibial osteotomy or femoral osteotomy.
* Patients with neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* Patients with a systemic or metabolic disorder leading to progressive bone deterioration.
* Patients that are immunologically compromised, or receiving chronic steroids (>30 days), excluding inhalers.
* Patients bone stock is compromised by disease or infection, which cannot provide adequate support and/or fixation to the prosthesis.
* Patients with knee fusion to the affected joint.
* Patients with an active or suspected latent infection in or about the knee joint.
* Patients that are prisoners.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Internal database of prior total knee replacement patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Measurement of antero-posterior stability of the knee with stress x-rays. | 1 year post-operative
  Antero-posterior stability of the knee will be measured with stress x-rays using the TELOS Stress device in 45° and 90° flexion. Stress x-rays will be obtained during a single visit for subjects 1 year or greater post-operatively.

SECONDARY OUTCOMES:
Knee Society Score (KSS) | 1 year post-operative
  Clinical outcomes will be evaluated via the Knee Society Score (KSS) obtained during a single visit for subjects 1 year or greater post-operatively. The KSS is subdivided into a Knee Assessment score which rates only the knee joint itself, and a Functional Assessment score which rates the subject's ability to walk and climb stairs. Both scores range from 0-100, with a higher score indicating a better outcome.
Lower Extremity Activity Scale (LEAS) | 1 year post-operative
  Clinical outcomes will be evaluated via the Lower Extremity Activity Scale (LEAS) obtained during a single visit for subjects 1 year or greater post-operatively. The LEAS scale range is 1-18, with a higher value indicating a higher level of activity.
Forgotten Joint Score (FJS) | 1 year post-operative
  Clinical outcomes will be evaluated via the Forgotten Joint Score (FJS) obtained during a single visit for subjects 1 year or greater post-operatively. The FJS total score range is 0-100, with higher scores indicating a higher degree of "forgetting" the artificial joint, that is, a lower degree of awareness.

CONTACTS AND LOCATIONS:
Overall Officials: David F Scott, MD, Principal Investigator — Spokane Joint Replacement Center
Locations (1):
- Spokane Joint Replacement Center, Spokane, Washington, United States